CLINICAL TRIAL: NCT01830387
Title: Comparative Study of Polymetric Clips (Hem-o-Lok) Versus Historical Endoscopic Staplers for Laparoscopic Appendectomy
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00041869
Record Dates: First submitted 2013-04-03; First posted 2013-04-12 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Appendicitis
Keywords: Polymetric Clips (Hem-o-Lok); Laparoscopic Appendectomy; Endoscopic Staplers
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Polymetric clips: The study team will prospectively enroll subjects with a diagnosis of appendicitis who are scheduled for laparoscopic appendectomy to have Hem-o-Lok® clips used for closure of the appendiceal stump. All subjects enrolled in the study will have their medical chart reviewed from consent to 30 days post operatively.
  Interventions: Device: Polymetric clips
- Endoscopic Staplers: The study team will retrospectively identify patients who have undergone laparoscopic appendectomy during a one year time span by performing a database search. The operative notes will be reviewed for these patients to select patients who underwent ligation of the appendix with an endoscopic stapler.
  Interventions: Other: Endoscopic Staplers

INTERVENTIONS:
Device: Polymetric clips — The study team will prospectively enroll subjects with a diagnosis of appendicitis who are scheduled for laparoscopic appendectomy to have Hem-o-Lok® clips used for closure of the appendiceal stump.
  Groups: Polymetric clips
Other: Endoscopic Staplers — The study team will retrospectively identify patients who have undergone laparoscopic appendectomy by performing a database search. The operative notes will be reviewed for these patients to select patients who underwent ligation of the appendix with an endoscopic stapler.
  Groups: Endoscopic Staplers

SUMMARY:
The purpose of this study is to compare the clinical outcomes and the operative costs of appendectomy performed with the Hem-O-Lok polymetric clips compared to endoscopic staplers. Prospective data will be collected before, during, and after surgery on patients undergoing a laparoscopic appendectomy that have the Hem-o-Lok ® stapler used to close the stump after the appendix is removed. Use of the Hem-o-Lok ® stapler is standard for appendectomy patients at Duke Regional Hospital. Retrospective data will be collected from patients who had an appendectomy prior to 1/2012 using a different clip as part of their surgery, or an open appendectomy to compare outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. scheduled to undergo a laparoscopic appendectomy because of a diagnosis of appendicitis based on clinical history or radiographic imaging.

Exclusion Criteria:

1. Less than 18 years of age
2. Signs of appendiceal rupture or abcess on preoperative imaging studies (CT or ultrasound)
3. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged 18 years of age or older, scheduled to undergo a laparoscopic appendectomy because of a diagnosis of appendicitis based on clinical history or radiographic imaging.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Length of stay | Subjects will be followed for the duration of their hopsital stay, an expected average of 2-3 days.
  Charts will be reviewed to calculate the number of days the subject was in the hospital. Clinical and financial outcomes of subjects enrolled for laparoscopic appendectomy using Hem-o-Lok will be compared to a historical (retrospective) cohort of patients who underwent appendectomy using endoscopic staplers.
Total Hospital Charges | Financial data will be gathered for the duration of the subjects hospital stay, an expected average of 2-3 days.
  Data will be gathered on the expense of the subjects hospital stay from admission, surgery, to discharge. Clinical and financial outcomes of subjects enrolled for laparoscopic appendectomy using Hem-o-Lok will be compared to a historical (retrospective) cohort of patients who underwent appendectomy using endoscopic staplers.
Operative time | Length of operation is approximately one and a half hours
  Subject's chart will be reviewed to gather operative start and stop times. Clinical and financial outcomes of subjects enrolled for laparoscopic appendectomy using Hem-o-Lok will be compared to a historical (retrospective) cohort of patients who underwent appendectomy using endoscopic staplers.

SECONDARY OUTCOMES:
Rates of Surgical Outcomes | Immediatly Postoperative to 30 days postoperative
  Measures of surgical outcomes will be compared between the two procedures including rates of postoperative appendiceal stump dehiscence, hemorrhage, pneumonia, urinary tract infection, myocardial infarction, pulmonary embolism, deep vein thrombosis, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Chan Park, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Metabolic and Weight Loss Surgery, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No